CLINICAL TRIAL: NCT00002068
Title: A Multicenter Comparison of Fluconazole (UK-49,858) and Amphotericin B as Treatment for Acute Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012H; 056-159B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Drug Therapy, Combination; Fluconazole; Flucytosine; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety and effectiveness of fluconazole and amphotericin B, alone or in combination with flucytosine, as treatment for acute cryptococcal meningitis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Written informed consent must be obtained for each patient, either from the patient himself or from the patient's legal guardian.

* No prior systemic antifungal therapy for cryptococcosis.
* Relapse after prior therapy.
* Success of prior therapy must have been documented by negative cerebrospinal fluid (CSF) culture at the end of therapy. Following prior therapy, such patients may not have received more than 1 mg/kg/wk amphotericin B in the 4 weeks before entry into study.

Prior Medication:

Allowed:

* Immunosuppressant therapy.
* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.
* Comatose.
* Unlikely to survive more than 2 weeks.

Concurrent Medication:

Excluded within 4 weeks of study entry:

* Greater than 1 mg/kg/wk amphotericin B.
* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.
* Comatose.
* Unlikely to survive more than 2 weeks.

Prior Medication:

Excluded within 4 weeks of study entry:

* Greater than 1 mg/kg/wk amphotericin B.
* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Davies Med Ctr, San Francisco, California
  - Christiana Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Univ of South Florida, Tampa, Florida
  - Univ of Maryland / Inst of Human Virology, Baltimore, Maryland
  - Henry Ford Hosp, Detroit, Michigan
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Univ of Tennessee, Memphis, Tennessee
- Saint Michael's Hosp, Toronto, Ontario, Canada